CLINICAL TRIAL: NCT01233310
Title: Evaluation of Small Bowel Colon Capsule for Bowel Visualization in Crohn's Disease Patients
Acronym: SBC-CD
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: RD-302
Record Dates: First submitted 2010-11-01; First posted 2010-11-03 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2012-08

CONDITIONS: Crohn Disease
Keywords: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Study Hypothesis:

It is estimated that by re-programming some of the PillCam COLON2 system parameters it can serve as tool for visualizing both small bowel and colon. As such, the system may be utilized in CD patients for monitoring mucosal healing.

Primary objectives:

To evaluate two different video output methods in the visualization of the SB and colon in CD patients

Secondary objectives:

* Evaluate the level of agreement between PillCam system and ileocolonoscopy on the assessment of CD findings.
* Evaluate the effectiveness of PillCam regimen in CD patients

Inclusion criteria

* Patient is 18 years of age and above
* Patient with a diagnosis of ileocolonic or colonic Crohn's Disease documented by endoscopical, histopathological and/or radiological parameters
* Patients' CDAI >150.
* Patient is clinically indicated to undergo ileocolonoscopy for assessment of Crohn's disease
* Proven patency by Agile capsule or another approach deemed clinically acceptable by the investigator, e.g. CT enterography, performed within the 3 months prior to enrollment
* Patient is able and agrees to sign the Informed Consent Form

Exclusion criteria

* Patient has dysphagia
* Patient has congestive heart failure
* Patient has renal insufficiency
* Patient has cirrhosis
* Patient is known or is suspected to suffer from intestinal obstruction
* Patient has known previous stricture/obstruction of the SB or colon
* Patient has taken NSAID medications less than one month before enrollment
* Patient suffers from hypertension and is taking one or more of the following medications used for control of hypertension: diuretics, ACE inhibitors, Angiotensin II blockers
* Chronic use of laxatives
* Patient has a cardiac pacemakers or other implanted electro medical devices.
* Women who are either pregnant or nursing at the time of screening, who intend to be during the study period, or are of child-bearing potential and do not practice medically acceptable methods of contraception.
* Patient is expected to undergo MRI examination within 7 days after ingestion of the capsule.
* Patient has had prior abdominal surgery of the gastrointestinal tract other than uncomplicated procedures that would be unlikely to lead to bowel obstruction based on the clinical judgment of the investigator.
* Patient has any condition, which precludes compliance with study and/or device instructions.
* Patient suffers from life threatening conditions
* Patient is currently participating in another clinical study
* Patient has known slow gastric emptying time
* Patient is allergic or contraindicated to any of the study medications

DETAILED DESCRIPTION:
Study design: Multi-center, prospective study Number of subjects: Up to 30 study duration: up to 18 months Subject population: Subjects with moderate to severe Crohn's disease demonstrating colon involvement who are indicated to undergo standard ileocolonoscopy as part of their disease management

Study Design:

1. Each patient will undergo PillCam, procedure followed by conventional ileocolonoscopy procedure with intubation of the terminal ileum
2. During the ileocolonoscopy procedure, the colonoscopist will document his findings according to the parameters defined in the SES-CD score and the overall assessment in the following segments:

   1. Rectum
   2. Left colon (including sigmoid)
   3. Transverse colon
   4. Right colon
   5. Terminal ileum
3. Cleansing level for the ileocolonoscopy procedure will be assessed at each site
4. From each capsule endoscopy procedure two RAPID video versions will be generated and segmented into segments
5. A committee composed of the study investigators will review all the RAPID video segments and document their findings according to the parameters defined in the SES-CD, Lewis and CECDAI scoring systems and an overall assessment
6. The parameters for each segment per each of the two RAPID movies will be compared and the preferable video setup will be chosen
7. Final RAPID and colonoscopy movies will be de-identified in regards to patient and site identity
8. The preferable full RAPID version will be reviewed by investigators which will document their findings according to the parameters defined in the SES-CD scoring system and overall assessment
9. cleansing level for the capsule procedure will be assess

The above evaluations per each subject will be within 24 from end of rocedure.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years of age and above
* Patient with a diagnosis of ileocolonic or colonic Crohn's Disease documented by endoscopical, histopathological and/or radiological parameters
* Patients' CDAI >150.
* Patient is clinically indicated to undergo ileocolonoscopy for assessment of Crohn's disease
* Proven patency by Agile capsule or another approach deemed clinically acceptable by the investigator, e.g. CT enterography, performed within the 3 months prior to enrollment
* Patient is able and agrees to sign the Informed Consent Form

Exclusion Criteria:

* Patient has dysphagia
* Patient has congestive heart failure
* Patient has renal insufficiency
* Patient has cirrhosis
* Patient is known or is suspected to suffer from intestinal obstruction
* Patient has known previous stricture/obstruction of the SB or colon
* Patient has taken NSAID medications less than one month before enrollment
* Patient suffers from hypertension and is taking one or more of the following medications used for control of hypertension: diuretics, ACE inhibitors, Angiotensin II blockers
* Chronic use of laxatives
* Patient has a cardiac pacemakers or other implanted electro medical devices.
* Women who are either pregnant or nursing at the time of screening, who intend to be during the study period, or are of child-bearing potential and do not practice medically acceptable methods of contraception.
* Patient is expected to undergo MRI examination within 7 days after ingestion of the capsule.
* Patient has had prior abdominal surgery of the gastrointestinal tract other than uncomplicated procedures that would be unlikely to lead to bowel obstruction based on the clinical judgment of the investigator.
* Patient has any condition, which precludes compliance with study and/or device instructions.
* Patient suffers from life threatening conditions
* Patient is currently participating in another clinical study
* Patient has known slow gastric emptying time
* Patient is allergic or contraindicated to any of the study medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Crohn's disease clinic
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2010-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Agreement level between two PillCam videos, simulating different proposed system setups, on the severity and extent of CD lesions,up to 24 months | up to 24 months

SECONDARY OUTCOMES:
Agreement level between PillCam and conventional ileocolonoscopy on the severity and extent of CD lesions, at colon and terminal ileum, based on the SES-CD score parameters and an overall assessment per each segment, up to 24 months | up to 24 months
Capsule transit time statistics within stomach, small bowel and colon segments,up to 24 months | up to 24 months
Capsule excretion time statistics, up to 24 months | up to 24 months
Assessment of colon and SB cleansing level at different colon and SB,up to 24 months | up to 24 months
Number, type and severity of adverse events, up to 24 months | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Niv, Professor, Principal Investigator — Belinson medical center; Abraham Eliakim, Professor, Principal Investigator — Rambam Health Care center
Locations (4):
- Israel (4):
  - Rambam Health Care center, Haifa
  - Bikur Holim medical center, Jerusalem
  - Belinson medical center, Petah Tikva
  - Asaf Harofe medical center, Zrifin